CLINICAL TRIAL: NCT03034811
Title: Persona Partial Knee Clinical Outcomes Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K.CR.I.G.16.16
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis; Avascular Necrosis; Traumatic Arthritis; Conditional Tibial Condyle or Plateau Fractures; Conditional Revision of the Articular Surface
Keywords: Noninflammatory degenerative joint disease; Osteoarthritis; Avascular necrosis; Traumatic arthritis; Partial knee arthroplasty; Unicompartmental knee arthroplasty
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PPK subjects (Other): Subjects that receive the Persona Partial Knee system
  Interventions: Device: Persona Partial Knee system

INTERVENTIONS:
Device: Persona Partial Knee system — Fixed bearing partial knee

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcomes data for the commercially available Persona Partial Knee System.

DETAILED DESCRIPTION:
The study design is a prospective, multicenter, noncontrolled study of the commercially available Persona Partial Knee. The study will require each site to obtain IRB approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their partial knee arthroplasty. Investigators will collect clinical data for a required 2 years with the option to continue follow-up assessment up to 10 years. Follow-up clinical visits include 3 months, 1 year, 2, 5, and 10 years post-operatively.

The primary objective of this study is to obtain implant survivorship and clinical outcomes data for the commercially available Persona Partial Knee System. The assessments will include: implant survivorship based on revision with removal of the study device; safety based on incidence and frequency of adverse events; and clinical performance measured by overall pain and function, quality of life data, radiographic parameters, and survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient qualifies for knee arthroplasty based upon physical exam and medical history, and meets the approved indications for use of the Persona Partial Knee system.
* Patient has participated in a study-related Informed Consent process
* Patient is willing and able to provide written Informed Consent by signing and dating the IRB/EC approved Informed Consent form
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations
* Independent of study participation, patient is a candidate for the commercially available Persona Partial Knee, implanted in accordance with product labeling

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies
* Infection, sepsis, and osteomyelitis
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Insufficiency of the collateral, anterior or posterior cruciate ligaments which would preclude stability of the device
* Full thickness damage to the weight bearing area of the contralateral compartment
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Insufficient bone stock to provide adequate support and/or fixation to the prosthesis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee
* Charcot's disease
* Fixed varus deformity (not passively correctable) of greater than 15 degrees
* Fixed flexion deformity (not passively correctable) of greater than 15 degrees
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score | 10 years
  A Patient reported functional outcome score for knee arthroplasty

SECONDARY OUTCOMES:
EQ-5D | 10 years
  a questionnaire completed by the Patient and assesses his/her General health Status. The EQ5D is used to derive a Quality of life index used for health economics considerations.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (24):
- United States (9):
  - Sah Orthopaedic Associates, Fremont, California
  - Panorama Orthopedics & Spine Center, Golden, Colorado
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Henry County Orthopedics and Sports Medicine, New Castle, Indiana
  - Sports Medicine North, Beverly, Massachusetts
  - Troy Orthopaedic Associates, Troy, Michigan
  - New Mexico Orthopaedics, Albuquerque, New Mexico
  - Midlands Orthopaedics & Neurosurgery, Columbia, South Carolina
  - Skagit Regional Clinics-Riverbend, Mount Vernon, Washington
- Orthopädisches Spital Speising, Vienna, Austria
- Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Belgium
- France (2):
  - Marseille University-Hospital Centres, Marseille
  - Public Hospital of Versailles, Versailles
- Germany (3):
  - Hessing Stiftung, Augsburg
  - Sana Kliniken Sommerfeld, Berlin
  - Waldkrankenhaus Eisenberg, Eisenberg
- Italy (2):
  - Orthopedic Institute IRCCS, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Hospital Alcorcón, Madrid, Spain
- Umea University Hospital, Umeå, Sweden
- Hopital d'Yverdon les Bains, Yverdon-les-Bains, Switzerland
- United Kingdom (3):
  - Avon Orthopaedic Centre, Southmead Hospital, Bristol
  - Royal Derby Hospital, Derby
  - Harrogate and District NHS Foundation Trust, Harrogate

IPD SHARING:
Plan to Share IPD: No